CLINICAL TRIAL: NCT02007096
Title: Transabdominal Plane (TAP) Blocks in Ventral Hernia Repair
Brief Title: Does a Transabdominal Plane Block Decrease Patient Pain After Ventral Hernia Repair?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Celia M. Divino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GCO 12-0960
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Ventral Hernia; Umbilical Hernia; Incisional Hernia; Postoperative Complications; Pain, Postoperative
Keywords: Transabdominal plane block; ventral hernia; umbilical hernia; incisional hernia; hernia repair
MeSH Terms: conditions — Hernia, Ventral; Hernia, Umbilical; Incisional Hernia; Postoperative Complications; Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transabdominal Plane Block (Experimental): Receiving Transabdominal Plane Block with 0.25% bupivacaine
  Interventions: Drug: Transabdominal Plane Block
- Non Transabdominal Plane Block (Placebo Comparator): Receiving placebo saline injection
  Interventions: Drug: Non Transabdominal Plane Block

INTERVENTIONS:
Drug: Transabdominal Plane Block — 0.25% bupivacaine injection in 6 different locations in abdomen. Weight <100kg: 50ml total; weight >100kg: 60ml total
  Other Names: Bupivacaine
  Arms: Transabdominal Plane Block
Drug: Non Transabdominal Plane Block — Saline injection in 6 different locations in abdomen. Weight <100kg: 50ml; weight >100kg: 60ml
  Other Names: Saline
  Arms: Non Transabdominal Plane Block

SUMMARY:
The purpose of this study is to determine if a Transabdominal Plane Block will decrease patient pain and pain medication use after a laparoscopic ventral (ventral, umbilical, incisional) hernia repair with mesh.

DETAILED DESCRIPTION:
Patients coming in for a laparoscopic ventral (ventral, umbilical, incisional) hernia repair with mesh are randomized to either receive a Transabdominal Plane Block injection or a placebo saline injection. The injection will be performed by surgeons under direct visualization during laparoscopic surgery prior to mesh placement. Patients will be followed up post-operatively and after hospital discharge to assess for opioid usage and pain score. Patients in both arms are medically cleared by the surgeon. Currently there are no studies that look at the use of Transabdominal Plane Block in ventral hernia repairs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* elective laparoscopic ventral (ventral, umbilical, incisional) hernia repair at Mount Sinai Hospital

Exclusion Criteria:

* age younger than 18
* allergic reaction to bupivacaine
* allergic reaction to opioids
* opioid substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celia M Divino, MD, FACS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Fields AC, Gonzalez DO, Chin EH, Nguyen SQ, Zhang LP, Divino CM. Laparoscopic-Assisted Transversus Abdominis Plane Block for Postoperative Pain Control in Laparoscopic Ventral Hernia Repair: A Randomized Controlled Trial. J Am Coll Surg. 2015 Aug;221(2):462-9. doi: 10.1016/j.jamcollsurg.2015.04.007. Epub 2015 Apr 22. PMID 26206644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the Department of Surgery at The Mount Sinai Hospital between November 2012 and October 2014.
Groups:
- Transabdominal Plane Block: Transabdominal Plane Block with 0.25% bupivacaine
- Non Transabdominal Plane Block: Non Transabdominal Plane Block: Saline injection
Period: Overall Study
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block
Started | 63 | 64
Completed | 52 | 48
Not Completed | 11 | 16
Not completed — medication not available | 2 | 0
Not completed — did not inject saline | 0 | 3
Not completed — did not follow postoperative protocol | 8 | 11
Not completed — converted to open surgery | 1 | 1
Not completed — no mesh placed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.67 (12.89) | 53.81 (13.45) | 53.22 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 25 | 27 | 52
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 30.91 (5.45) | 31.16 (7.00) | 31.03 (6.21)
ASA class [Count of Participants; unit: Participants] — Preoperative American Society of Anesthesia (ASA) scores to evaluate the degree of a patient's "sickness" or "physical state" before selecting the anesthetic or before performing surgery, with one being normal to five being severely impaired.
  Participants
    1 | 7 | 6 | 13
    2 | 24 | 24 | 48
    3 | 20 | 16 | 36
    4 | 1 | 2 | 3
Hypertension [Count of Participants; unit: Participants] | 25 | 23 | 48
Diabetes [Count of Participants; unit: Participants] | 10 | 9 | 19
Hyperlipidemia [Count of Participants; unit: Participants] | 14 | 20 | 34
Coronary artery disease [Count of Participants; unit: Participants] | 6 | 9 | 15
GERD [Count of Participants; unit: Participants] — Gastroesophageal reflux disease
  Participants | 12 | 13 | 25
Smoker [Count of Participants; unit: Participants] | 15 | 17 | 32
Previous abdominal surgery [Count of Participants; unit: Participants] | 41 | 31 | 72
Hernia defect size [Mean (Standard Deviation); unit: cm^2] | 38.46 (42.26) | 39.84 (61.27) | 39.12 (51.99)
Location of hernia defect [Count of Participants; unit: Participants]
  Epigastric | 23 | 18 | 41
  Umbilical | 19 | 20 | 39
  Infraumbilical | 2 | 7 | 9
  Lateral | 8 | 3 | 11
LOS [Count of Participants; unit: Participants] — length of stay
  Participants
    <2 days | 35 | 36 | 71
    ≥2 days | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Use
Description: Amount of opioids used by patients at certain time points.
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block
Number analyzed (Participants) | 52 | 48
mg
  at 6 hours | 10.59 (0) | 15.62 (0)
  at 12 hours | 16.09 (0) | 32.24 (0)
  at 18 hours | 20.70 (0) | 39.37 (0)
  at 24 hours | 25.64 (0) | 42.56 (0)

2. Secondary Outcome: Pain Score
Description: Post-operative Patient Self-Reported Pain Score. Patient self-reported pain scores when resting and when actively moving. Scale of 0 to 10, with 0 being "no pain" and 10 being "the most pain you have ever experienced."
Time Frame: 1 hour postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block
Number analyzed (Participants) | 52 | 48
units on a scale
  pain scores at rest | 5.19 (0.39) | 6.46 (0.38)
  pain scores with movement | 6.15 (0.42) | 7.73 (0.40)

3. Secondary Outcome: Operating Procedure Time
Description: Total number of minutes for the procedure, not including anesthesia time.
Time Frame: Procedure begin time to procedure end time
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block
Number analyzed (Participants) | 52 | 48
min | 97.41 (30.22) | 98.81 (37.51)

4. Secondary Outcome: Pain Score
Description: as for outcome 2
Time Frame: 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block
Number analyzed (Participants) | 52 | 48
units on a scale
  pain scores at rest | 4.60 (0.39) | 4.52 (0.31)
  pain scores with movement | 6.75 (0.38) | 6.98 (0.40)

ADVERSE EVENTS:
Description: Adverse Events information not collected
Arm/Group | Transabdominal Plane Block | Non Transabdominal Plane Block
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The surgeon knew the group assignment to administer the correct injection. Data not collected on clinical difference, e.g. postop nausea & vomiting. Study conducted at one center with experienced surgeons, so the results might not be generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes